CLINICAL TRIAL: NCT01193582
Title: A Phase 4, Open-label Trial to Assess the Safety, Tolerability and Immunogenicity of Prevenar in Older Infants and Young Children in China Who Are Naive to Previous Pneumococcal Vaccination.
Brief Title: A Study To Assess The Safety And Effectiveness Of Prevenar In Chinese Children Who Have Not Previously Received A Vaccine Against Pneumococcal Bacteria
Acronym: 6114A1-4000-CN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B1841008; B1841008
Record Dates: First submitted 2010-08-31; First posted 2010-09-02 (Estimated); Results first posted 2013-11-20 (Estimated); Last update posted 2013-11-20 (Estimated); Status verified 2013-09

CONDITIONS: Pneumococcal Infections
Keywords: Prevenar; catch-up; pneumococcal; pneumonia
MeSH Terms: conditions — Pneumococcal Infections; Pneumonia | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group 1 (Experimental)
  Interventions: Biological: Prevenar
- Group 2 (Experimental)
  Interventions: Biological: Prevenar
- Group 3 (Experimental)
  Interventions: Biological: Prevenar
- Group 4 (Experimental)
  Interventions: Biological: Prevenar

INTERVENTIONS:
Biological: Prevenar — Dosage form: intramuscular injection Dosage: 0.5 ml
  Frequency:
  4 doses starting from 121 to < 212 days of age
  Arms: Group 1
Biological: Prevenar — Dosage form: intramuscular injection Dosage: 0.5 ml
  Frequency:
  3 doses starting from 212 days to < 12 months of age
  Arms: Group 2
Biological: Prevenar — Dosage form: intramuscular injection Dosage: 0.5 ml
  Frequency:
  2 doses starting from 12 months to < 24 months of age
  Arms: Group 3
Biological: Prevenar — Dosage form: intramuscular injection Dosage: 0.5 ml
  Frequency:
  1 dose starting from 24 months to < 72 months of age
  Arms: Group 4

SUMMARY:
A vaccine called Prevenar is already approved for use in China for vaccination of children younger than 6 years old against infections caused by Streptococcus pneumoniae.

This study is to measure the amount of antibodies (antibodies help people fight off diseases) Chinese children aged between 121 days and 6 years (72 months) produce when given Prevenar. The study will also provide more data on how safe and well tolerated Prevenar is in Chinese children.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Chinese male or female subjects.
* Between 121 days to less than 72 months of age at the time of entry into the study.

Exclusion Criteria:

* Receipt of previous vaccine against Pneumo
* Previous anaphylactic reaction to any vaccine or part of a vaccine
* Previous proven invasive Pneumo infection
* Receipt of investigational drug or device within the proceeding 28 days

Ages: 121 Days to 72 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 505 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- China (5):
  - Baolixiang Clinic, Baoli Town,Yongfu County, Guangxi
  - Guangfuxiang Clinic, Guangfu Town, Yongfu County, Guangxi
  - Luojin Clinic, Luojin Town, Yongfu County, Guangxi
  - Yongfu County CDC, Yongfu County, Guangxi
  - Yongfu County Clinic, Yongfu County, Guangxi

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1841008&StudyName=A%20Study%20To%20Assess%20The%20Safety%20And%20Effectiveness%20Of%20Prevenar%20In%20Chinese%20Children%20Who%20Have%20Not%20Previously%20Received%20A%20Vaccine%20Against%20Pn

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This report presents results following completion of all vaccinations, including data from the 12-month follow-up. This study was conducted at one site in China.
Pre-assignment Details: Participants were enrolled into 1 of 4 groups based on inclusion/exclusion criteria without a screening period.
Groups:
- Group 1: Participants 121 to <212 days of age and received 4 doses of Prevenar.
- Group 2: Participants 212 days to <12 months of age (before the first birthday) and received 3 doses of Prevenar.
- Group 3: Participants 12 to <24 months of age (before the second birthday) and received 2 doses of Prevenar
- Group 4: Participants 24 to <72 months of age (before the sixth birthday) and received 1 dose of Prevenar
Period: Vaccination Series
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 100 | 101 | 125 | 180
Vaccinated Dose 1 | 100 | 100 | 125 | 180
Vaccinated Dose 2 | 92 | 91 | 118 | 0
Vaccinated Dose 3 | 90 | 89 | 0 | 0
Vaccinated Dose 4 | 90 | 0 | 0 | 0
Completed | 89 | 88 | 117 | 177
Not Completed | 11 | 13 | 8 | 3
Not completed — Withdrawal by Subject | 11 | 13 | 8 | 3
Period: 12 Month Follow-up
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 89 | 88 | 117 | 177
Completed | 83 | 88 | 113 | 166
Not Completed | 6 | 0 | 4 | 11
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 3 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 88 | 87 | 115 | 177 | 467
Age Continuous [Mean (Standard Deviation); unit: Months] — Age at first Vaccination
  Months | 5.3 (0.9) | 9.8 (1.4) | 17.5 (4.2) | 44.5 (13.0) | 24.0 (18.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 43 | 58 | 93 | 244
  Male | 38 | 44 | 57 | 84 | 223

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations to the 7 Pneumococcal Serotypes Contained in Prevenar
Description: Serotype-specific Pneumococcal Immunoglobulin G (IgG) antibody geometric mean concentration (GMC) after 1 month of last dose for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% confidence intervals (CI) were evaluated. Geometric means (GMs) were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after last dose in each group
Population: Evaluable immunogenicity population consisted of eligible participants in the age range who had received all the assigned vaccination(s), had blood drawn within required time frames, had at least 1 valid and determinate assay result for the proposed analysis, had received no prohibited vaccines, and had no other major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 100 | 101 | 125 | 180
μg/mL
  Serotype 4 (n= 88, 87, 115, 177) | 6.90 [5.61 to 8.48] | 7.16 [6.09 to 8.42] | 7.53 [6.70 to 8.46] | 9.45 [8.38 to 10.65]
  Serotype 6B (n= 88, 87, 114, 177) | 8.01 [6.24 to 10.30] | 5.79 [4.64 to 7.23] | 4.81 [3.89 to 5.96] | 6.36 [5.32 to 7.59]
  Serotype 9V (n= 88, 87, 115, 177) | 4.11 [3.40 to 4.96] | 4.64 [3.93 to 5.47] | 4.67 [4.18 to 5.21] | 6.14 [5.42 to 6.95]
  Serotype 14 (n= 88, 87, 115, 177) | 12.75 [10.32 to 15.76] | 13.02 [10.89 to 15.57] | 11.98 [10.51 to 13.65] | 9.86 [8.03 to 12.10]
  Serotype 18C (n= 88, 87, 115, 177) | 4.65 [3.81 to 5.69] | 4.65 [3.86 to 5.61] | 5.40 [4.78 to 6.10] | 7.39 [6.41 to 8.51]
  Serotype 19F (n= 87, 87, 115, 177) | 4.05 [3.07 to 5.36] | 4.02 [3.05 to 5.31] | 4.03 [3.26 to 4.98] | 4.53 [3.73 to 5.49]
  Serotype 23F (n= 88, 87, 115, 177) | 4.75 [3.77 to 5.99] | 3.95 [3.19 to 4.89] | 4.18 [3.51 to 4.96] | 5.64 [4.84 to 6.57]

2. Primary Outcome: Antibody Concentrations to the 7 Pneumococcal Serotypes Contained in Prevenar at Baseline in Each Group
Description: Serotype-specific Pneumococcal IgG antibody GMC at baseline for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: Baseline
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 100 | 101 | 125 | 180
μg/mL
  Serotype 4 (n= 88, 87, 115, 172) | 0.01 [0.01 to 0.02] | 0.01 [0.01 to 0.02] | 0.02 [0.01 to 0.02] | 0.06 [0.05 to 0.08]
  Serotype 6B (n= 86, 64, 100, 177) | 0.12 [0.10 to 0.15] | 0.16 [0.12 to 0.22] | 0.27 [0.21 to 0.35] | 1.30 [1.08 to 1.55]
  Serotype 9V (n= 88, 84, 113, 177) | 0.10 [0.08 to 0.12] | 0.10 [0.08 to 0.13] | 0.17 [0.13 to 0.21] | 0.66 [0.56 to 0.77]
  Serotype 14 (n= 88, 87, 115, 177) | 0.16 [0.12 to 0.22] | 0.04 [0.03 to 0.05] | 0.03 [0.02 to 0.04] | 0.36 [0.26 to 0.50]
  Serotype 18C (n= 88, 87, 114, 172) | 0.04 [0.03 to 0.06] | 0.02 [0.01 to 0.02] | 0.02 [0.02 to 0.03] | 0.12 [0.10 to 0.16]
  Serotype 19F (n= 88, 85, 115, 169) | 0.11 [0.09 to 0.14] | 0.09 [0.07 to 0.12] | 0.13 [0.10 to 0.17] | 0.71 [0.57 to 0.89]
  Serotype 23F (n= 85, 75, 102, 174) | 0.07 [0.06 to 0.09] | 0.08 [0.06 to 0.11] | 0.17 [0.12 to 0.23] | 0.88 [0.74 to 1.04]

3. Secondary Outcome: Antibody Concentrations to the 7 Pneumococcal Serotypes Contained in Prevenar at 1 Month After the Third Dose in Group 1
Description: Serotype-specific Pneumococcal IgG antibody GMC one month after the third dose in Group 1 for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after third dose of Prevenar in Group 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 1
Number analyzed (Participants) | 100
μg/mL
  Serotype 4 (n= 88) | 6.38 [5.56 to 7.33]
  Serotype 6B (n= 87) | 2.88 [2.33 to 3.56]
  Serotype 9V (n= 88) | 4.18 [3.51 to 4.98]
  Serotype 14 (n= 88) | 11.16 [9.12 to 13.66]
  Serotype 18C (n= 88) | 4.60 [3.80 to 5.57]
  Serotype 19F (n= 88) | 3.60 [2.75 to 4.72]
  Serotype 23F (n= 88) | 2.45 [1.97 to 3.04]

4. Secondary Outcome: Geometric Mean Fold Rise (GMFR) of Anti-Pneumococcal Antibody Levels to the 7 Pneumococcal Serotypes Contained in Prevenar Above Vaccination Baseline Values in Group 1.
Description: GMFRs for the 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) from pre-vaccination to post-vaccination were computed using the logarithmically transformed assay results. CIs for GMFR are back transformations of a CI based on the Student t-distribution for the mean logarithm of the titers.
Time Frame: Pre-vaccination to 1 month after third dose of Prevenar in Group 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Group 1
Number analyzed (Participants) | 100
Fold rise
  Serotype 4 (n= 88) | 453.17 [344.56 to 596.01]
  Serotype 6B (n= 85) | 23.10 [18.15 to 29.40]
  Serotype 9V (n= 88) | 43.38 [33.42 to 56.32]
  Serotype 14 (n= 88) | 69.90 [45.95 to 106.35]
  Serotype 18C (n= 88) | 106.74 [76.83 to 148.31]
  Serotype 19F (n= 88) | 32.52 [23.39 to 45.21]
  Serotype 23F (n= 85) | 34.01 [24.98 to 46.32]

5. Secondary Outcome: Antibody Concentrations to the 7 Pneumococcal Serotypes Contained in Prevenar at 1 Month After the Second Dose in Group 2
Description: Serotype-specific Pneumococcal IgG antibody GMC 1 month after the second dose in Group 2 for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after second dose of Prevenar in Group 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 2
Number analyzed (Participants) | 101
μg/mL
  Serotype 4 (n= 87) | 8.46 [7.36 to 9.72]
  Serotype 6B (n= 85) | 2.67 [2.06 to 3.46]
  Serotype 9V (n= 87) | 4.71 [3.91 to 5.66]
  Serotype 14 (n= 87) | 8.05 [6.71 to 9.68]
  Serotype 18C (n= 87) | 4.93 [4.00 to 6.08]
  Serotype 19F (n= 87) | 3.03 [2.27 to 4.04]
  Serotype 23F (n= 87) | 2.66 [2.10 to 3.37]

6. Secondary Outcome: GMFR of Anti-Pneumococcal Antibody Levels to the 7 Pneumococcal Serotypes Contained in Prevenar Above Vaccination Baseline Values in Group 2.
Description: as for outcome 4
Time Frame: Pre-vaccination to 1 month after second dose of Prevenar in Group 2
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Group 2
Number analyzed (Participants) | 101
Fold rise
  Serotype 4 (n= 87) | 705.95 [540.50 to 922.05]
  Serotype 6B (n= 63) | 16.64 [11.17 to 24.79]
  Serotype 9V (n= 84) | 44.72 [34.22 to 58.44]
  Serotype 14 (n= 87) | 217.21 [152.52 to 309.33]
  Serotype 18C (n= 87) | 317.90 [219.65 to 460.10]
  Serotype 19F (n= 85) | 33.66 [24.28 to 46.65]
  Serotype 23F (n= 75) | 30.77 [21.30 to 44.45]

7. Secondary Outcome: Antibody Concentrations to the 7 Pneumococcal Serotypes Contained in Prevenar at 1 Month After the First Dose in Group 3
Description: Serotype-specific Pneumococcal IgG antibody GMC one month after the first dose in Group 3 for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 1 month after first dose of Prevenar in Group 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 3
Number analyzed (Participants) | 125
μg/mL
  Serotype 4 (n= 115) | 8.44 [7.25 to 9.81]
  Serotype 6B (n= 113) | 1.92 [1.51 to 2.42]
  Serotype 9V (n= 115) | 4.77 [4.09 to 5.56]
  Serotype 14 (n= 115) | 3.37 [2.74 to 4.16]
  Serotype 18C (n= 115) | 5.72 [4.82 to 6.77]
  Serotype 19F (n= 113) | 1.96 [1.55 to 2.49]
  Serotype 23F (n= 115) | 2.83 [2.26 to 3.53]

8. Secondary Outcome: GMFR of Anti-Pneumococcal Antibody Levels to the 7 Pneumococcal Serotypes Contained in Prevenar Above Vaccination Baseline Values in Group 3.
Description: as for outcome 4
Time Frame: Pre-vaccination to 1 month after first dose of Prevenar in Group 3
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Group 3
Number analyzed (Participants) | 125
Fold rise
  Serotype 4 (n= 115) | 476.49 [363.31 to 624.93]
  Serotype 6B (n= 99) | 7.06 [5.50 to 9.05]
  Serotype 9V (n= 113) | 28.11 [22.18 to 35.63]
  Serotype 14 (n= 115) | 108.18 [78.76 to 148.60]
  Serotype 18C (n= 114) | 236.39 [182.65 to 305.93]
  Serotype 19F (n= 113) | 15.13 [11.02 to 20.77]
  Serotype 23F (n= 102) | 17.64 [13.43 to 23.17]

9. Secondary Outcome: Antibody Concentrations Against the 7 Pneumococcal Serotypes Contained in Prevenar at 12 Months After the Last Dose.
Description: Serotype-specific Pneumococcal IgG antibody GMC 12 months after the last dose for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) are presented. GMC and corresponding 2-sided 95% CI were evaluated. GMs were calculated using all participants with available data for the specified blood draw.
Time Frame: 12 months after the last dose
Population: Evaluable immunogenicity population consisted subjects who had received all , assigned vaccination(s), had blood drawn within required time frame for 12 month follow-up blood draw visit, had at least 1 valid and determinate assay result, had received no prohibited vaccines, and had no major protocol violations.
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 89 | 88 | 117 | 177
μg/mL
  Serotype 4 (n= 81, 79, 111, 162) | 0.78 [0.62 to 0.98] | 0.65 [0.52 to 0.82] | 0.96 [0.80 to 1.14] | 1.27 [1.11 to 1.45]
  Serotype 6B (n= 81, 78, 109, 161) | 3.22 [2.41 to 4.29] | 2.31 [1.77 to 3.03] | 2.38 [1.89 to 3.00] | 4.20 [3.49 to 5.04]
  Serotype 9V (n= 81, 79, 111, 162) | 1.26 [1.00 to 1.59] | 0.98 [0.79 to 1.21] | 1.44 [1.20 to 1.71] | 2.23 [1.94 to 2.56]
  Serotype 14 (n= 81, 79, 111, 162) | 1.84 [1.40 to 2.41] | 2.18 [1.62 to 2.94] | 2.61 [2.09 to 3.27] | 5.19 [4.25 to 6.33]
  Serotype 18C (n= 81, 79, 111, 162) | 0.87 [0.69 to 1.10] | 0.71 [0.59 to 0.85] | 0.98 [0.84 to 1.15] | 1.46 [1.24 to 1.72]
  Serotype 19F (n= 80, 76, 109, 156) | 1.25 [0.95 to 1.64] | 1.29 [0.85 to 1.95] | 1.39 [1.03 to 1.88] | 2.85 [2.28 to 3.56]
  Serotype 23F (n= 81, 78, 110, 162) | 1.38 [1.07 to 1.77] | 1.20 [0.91 to 1.59] | 1.79 [1.45 to 2.21] | 2.49 [2.13 to 2.92]

10. Secondary Outcome: GMFR of Anti-Pneumococcal Antibody Levels to the 7 Pneumococcal Serotypes Contained in Prevenar Above Vaccination Baseline Values at 12 Months After the Last Dose.
Description: GMFRs for the 7 pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) from pre-vaccination to 12- month follow-up were computed using the logarithmically transformed assay results. CIs for GMFR are back transformations of a CI based on the Student t-distribution for the mean logarithm of the titers.
Time Frame: Pre-vaccination to 12 months after the last dose
Population: as for outcome 9
Measure: Geometric Mean (95% Confidence Interval); unit: Fold rise
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 89 | 88 | 117 | 177
Fold rise
  Serotype 4 (n= 81, 79, 111, 157) | 52.86 [37.61 to 74.31] | 50.54 [37.47 to 68.18] | 52.19 [39.75 to 68.53] | 21.01 [17.04 to 25.91]
  Serotype 6B (n= 79, 58, 95, 161) | 25.52 [18.57 to 35.07] | 15.58 [10.18 to 23.83] | 7.99 [5.98 to 10.67] | 3.16 [2.70 to 3.70]
  Serotype 9V (n= 81, 76, 109, 162) | 12.73 [9.41 to 17.24] | 8.97 [6.84 to 11.77] | 8.40 [6.55 to 10.77] | 3.35 [2.93 to 3.83]
  Serotype 14 (n= 81, 79, 111, 162) | 10.19 [6.84 to 15.19] | 55.55 [37.23 to 82.87] | 88.27 [63.53 to 122.63] | 15.67 [11.43 to 21.47]
  Serotype 18C (n= 81, 79, 110, 158) | 19.75 [14.00 to 27.87] | 45.07 [33.12 to 61.33] | 41.14 [32.18 to 52.59] | 11.43 [9.38 to 13.92]
  Serotype 19F (n= 80, 74, 109, 150) | 10.06 [6.85 to 14.77] | 12.62 [8.67 to 18.39] | 11.15 [7.87 to 15.80] | 4.19 [3.19 to 5.51]
  Serotype 23F (n= 79, 67, 97, 159) | 18.80 [13.26 to 26.66] | 13.50 [9.56 to 19.04] | 11.39 [8.31 to 15.61] | 2.86 [2.39 to 3.42]

ADVERSE EVENTS:
Time Frame: Baseline through 12 months following last dose of Prevenar
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 1/100 | 0/100 | 1/125 | 0/180
Other Adverse Events (participants affected / at risk) | 3/100 | 4/100 | 3/125 | 1/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=100) | Group 2 (N=100) | Group 3 (N=125) | Group 4 (N=180)
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastroenteritis shigella (Infections and infestations) | 0 | 0 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=100) | Group 2 (N=100) | Group 3 (N=125) | Group 4 (N=180)
Pyrexia (General disorders) | 2 | 4 | 1 | 1
Hypersensitivity (Infections and infestations) | 0 | 0 | 1 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.